CLINICAL TRIAL: NCT03097055
Title: Acupuncture Intervention to Improve Neurological Function and Anti-inflammatory Effect in Patients With Acute Ischemic Stroke (ANAIS)
Brief Title: Acupuncture Intervention to Improve Neurological Function and Anti-inflammatory Effect in Acute Ischemic Stroke (ANAIS)
Acronym: ANAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Tsai Chueh-Yi, Master Student, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH106-REC1-008
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Acute Ischemic Stroke; Acupuncture
Keywords: Stroke; Acupuncture; antiinflammatory; NIHSS
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Acupuncture (Experimental): Traditional acupoints and traditional "deqi" manipulation
  Interventions: Procedure: Traditional Acupuncture
- Minimal Acupuncture (Sham Comparator): To avoid traditional acupoints and minimal manipulation
  Interventions: Procedure: Minimal Acupuncture

INTERVENTIONS:
Procedure: Traditional Acupuncture — widely ongoing traditional acupoints in scalp and limbs with traditional "deqi" manipulation, for stroke patient
  Arms: Traditional Acupuncture
Procedure: Minimal Acupuncture — non-traditional acupoints in scalp and limbs, with minimal manipulation
  Arms: Minimal Acupuncture

SUMMARY:
This study will have acupuncture intervention in acute ischemic stroke patients and evaluate the effect in neurological function improving by National Institutes of Health Stroke Scale (NIHSS), Modified Rankin Scale (mRS), Barthel Index, and antiinflammatory actions by biomarkers.

DETAILED DESCRIPTION:
Acupuncture Treatment in Stroke is a widely practiced in Taiwan, mainland China, and around the world. The using in stroke group is countless. Numerous clinical trials have been conducted in the medical community to assess efficacy, and the results mostly suggest that acupuncture may be an effective, low side effects adjuvant therapy. Ischemic stroke is also associated with chronic inflammation-related diseases. In recent years, the anti-inflammatory effect of acupuncture was gradually found. So, whether in the basic or in clinical, the investigators can deduce that acupuncture may be helpful for stroke as an adjuvant therapy.

This study evaluates the neurological function of patients with acute stroke by using the widely used National Institutes of Health Stroke Scale (NIHSS), Modified Rankin Scale (mRS) and Barthel Index. Also, the investigators assess the degree of inflammation by biomarkers. Therefore, the purpose of this study is to explore the effect of acupuncture intervention on acute ischemic patients and its relationship in anti-inflammatory actions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed acute ischemic stroke
* Initial NIHSS between 4~20
* Aged 45 ~ 85

Exclusion Criteria:

* Hemorrhagic transformation after cerebral infarction, the hemorrhage size estimated to be ≥ 2cm in diameter by brain imaging.
* Any intracranial hemorrhage , except hemorrhagic transformation after cerebral infarction
* Any intracranial operation during acute stage
* Patient using anticoagulants
* Cerebellar infarction
* Special causes of stroke, such as coagulation abnormalities, or arteriovenous malformations
* Epileptic seizures after stroke
* Combined with infection diseases at the time of assessment
* Pregnant or breastfeeding women
* Present mental illness or symptoms and cannot cooperate with the study
* Cannot sign the inform consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 1.beginning of stroke (within 3 days after onset); 2.after a 4-weeks acupuncture course (within 7 days after last acupuncture); 3. a month later after acupuncture course (about 28±7 days after last acupuncture)
  The NIHSS improving in about a 2-months-period follow up.

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | 1.beginning of stroke (within 3 days after onset); 2.after a 4-weeks acupuncture course (within 7 days after last acupuncture); 3. a month later after acupuncture course (about 28±7 days after last acupuncture)
  The mRS improving in about a 2-months-period follow up.
Barthel Index | 1.beginning of stroke (within 3 days after onset); 2.after a 4-weeks acupuncture course (within 7 days after last acupuncture); 3. a month later after acupuncture course (about 28±7 days after last acupuncture)
  The Barthel Index improving in about a 2-months-period follow up.
inflammatory biomarkers | 1.beginning of stroke (within 3 days after onset); 2.after a 4-weeks acupuncture course (within 7 days after last acupuncture); 3. a month later after acupuncture course (about 28±7 days after last acupuncture)
  The inflammatory biomarkers changing in about a 2-months-period follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Yi Tsai, MD, Principal Investigator — Nantou Hospital of the Ministry of Health and Welfare, Taiwan; China Medical University, Taiwan; Ching-Liang Hsieh, MD/PhD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- Nantou Hospital of the Ministry of Health and Welfare, Nantou City, Nantou County, Taiwan

IPD SHARING:
Plan to Share IPD: No